CLINICAL TRIAL: NCT02213510
Title: A Prospective, Non-blinded, Randomized Controlled Post-market Study Designed to Compare the Use of the Zip Surgical Skin Closure Device Versus Conventional Sutures for Skin Closure in Subjects Who Undergo a CIED Procedure.
Brief Title: ZIPS Study - Zip Incision aPproximation vs. Suture
Acronym: ZIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: ZipLine Medical Inc. (Industry)
Responsible Party: Principal Investigator, Ulrika Birgersdotter-Green, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 140718
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Wound; Cardiac Arrhythmia
Keywords: pacemaker; implantable cardioverter defibrillator; ICD; surgical wound closure; sutures; Zipline; Zips; CIED; cardiovascular implantable electronic devices; arrhythmia
MeSH Terms: conditions — Wounds and Injuries; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zip Surgical Skin Closure device (Experimental): The Zip Surgical Skin Closure device is a single use, sterile medical device that replaces sutures, staples, and glue for closure of the skin layer for surgical incisions or laceration repair. The device will applied by the surgeon at the end of the CIED procedure and be worn until the two week post-operative wound check.
  Interventions: Device: Zip Surgical Skin Closure Device
- Standard Suture Closure (Active Comparator): The surgeon will perform standard suture closure for the skin layer following CIED procedure.
  Interventions: Device: Standard Suture Closure

INTERVENTIONS:
Device: Zip Surgical Skin Closure Device — The Zip Surgical Skin Closure device is a single use, sterile medical device that replaces sutures, staples, and glue for closure of the skin layer for surgical incisions or laceration repair. The device will applied by the surgeon at the end of the CIED procedure and be worn until the two week post-operative wound check.
  Other Names: Wound closure device
  Arms: Zip Surgical Skin Closure device
Device: Standard Suture Closure — The surgeon will perform standard suture closure for the skin layer following CIED procedure.
  Arms: Standard Suture Closure

SUMMARY:
ZipLine Medical, Inc. has developed a novel, non-invasive skin closure device called "Zip Surgical Skin Closure" to replace sutures, staples and glue for closure of the skin layer for surgical incisions or laceration repair. The study will be comparing the Zip Surgical Skin Closure to standard sutures in patients undergoing cardiovascular implantable electronic device (CIED) procedures on outcomes including closure time, cosmetic appearance of resulting scar, and overall cosmetic appearance of scar. The study will be following participants for 3 months following CIED procedure.

DETAILED DESCRIPTION:
ZipLine Medical, Inc. has developed a novel, non-invasive skin closure device called "Zip Surgical Skin Closure" to replace sutures, staples and glue for closure of the skin layer for surgical incisions or laceration repair. The device is designed to provide closure speed superior to sutures, while resulting in a suture-like cosmetic outcome.The ZIPS study is a randomized, clinical trial comparing outcomes of procedures that use the Zip Surgical Skin Closure device with the outcomes of procedures that use stitches. The Zip Surgical Skin Closure is not an investigational device and is currently used in hospital across the United States. The Zip Surgical Skin Closure is a non-invasive (in other words, does not pierce the skin or enter into the wound) device to hold skin closed while healing can occur. It adheres to the skin close to the incision and uses adjustable straps to hold the incision closed. It is typically worn on the skin for 7-14 days and is removed by peeling from the skin. Patients will be randomized to either Zip Surgical Skin Closure or sutures, in addition to dissolvable sutures for the deeper layers, for surgical procedures for cardiovascular implantable electronic devices (CIED) i.e. pacemakers or defibrillators. Both of these closure techniques are considered standard of care at this facility and are not themselves experimental. However, the goal of this experimental study is to see if there are any significant differences between the two closure methods, in a controlled study environment.

Since the Zip Surgical Skin Closure device is relatively new to the market, there is a limited amount of information available describing the experience of patients and doctors using the device. In this study, the investigators will be looking to compare the Zip Surgical Skin Closure and stitches methods for the time necessary for the surgeon to close the incision, cosmetic appearance of the resulting scar, and satisfaction of you and your surgeon. The investigators will also be monitoring both study groups for occurrence of any adverse (unfavorable) events. Patients will be followed for a total of 3 months for this study. All study visits align with standard of care follow up for post-implantation of CIED. Non-identifiable pictures will be obtained of the scar during follow up and both patients and surgeons will complete questionnaires indicating their experience and satisfaction with the either skin closure method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and older;
2. Patients requiring suture closure for epidermal closure (after placement of cardiac implantable electronic devices; including de novo and re implant generator changes);
3. Patients willing and able to complete study protocol
4. Life expectancy greater than 1 year

Exclusion Criteria:

1. Known bleeding disorder not caused by medication;
2. Known personal or family history of keloid formation or scar hypertrophy;
3. Known allergy or hypersensitivity to non-latex skin adhesives;
4. Atrophic skin deemed clinically prone to blistering;
5. Any skin disorder affecting wound healing;
6. Any other condition that in the opinion of the investigator would make a particular subject unsuitable for this study.
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Birgersdotter-Green, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

REFERENCES:
- See also: ZipLine Medical Website — http://www.ziplinemedical.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Started | 21 | 19
Completed | 20 | 18
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 71 [44 to 99] | 70 [41 to 100] | 70 [41 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
Fitzpatrick Skin Scale [Number; unit: participants]
  1 - Always burns, never tans | 2 | 0 | 2
  2 - Usually burns, tans with difficulty | 1 | 1 | 2
  3 - Somtimes mild burn, gradually tans | 7 | 6 | 13
  4 - Rarely burns, tans with ease | 6 | 7 | 13
  5 - Very rarely burns, tans very easily | 4 | 3 | 7
  6 - Never burns, tans very easily | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Closure Time
Description: Duration of time starting when suture needle (control) or Zip device touches the skin until final suture knot is cut or Zip device application is complete (e.g., top liner is removed.)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 19
seconds | 78 (30.36) | 216 (93.71)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Wound Healing as Determined by the CVAS (Cosmetic Visual Analogue Scale)
Description: Based on photographs taken of scars taken at 3 months following CIED procedure. The CVAS scale is measured from 0mm (representing best scar) to 100 mm (representing worst scar).
Time Frame: 3 Months
Population: Please note that only 18 patients were evaluated (of 19) in the Standard Suture Closure due to one patient withdrawing from the trial.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
mm | 35.8 (40.6) | 40.6 (21.7)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.655, t-test, 2 sided

3. Secondary Outcome: Surgeon Wound Evaluation Scale (WES)
Description: At 2 weeks post-procedure, the Wound Evaluation Scale was measured. The scale is based from 0 (representing normal skin) to 100 (representing a poor scar).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 19
units on a scale | 5.82 (0.50) | 5.78 (0.55)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.811, t-test, 2 sided

4. Secondary Outcome: Surgeon Evaluation Based on the Wound Evaluation Scale (WES)
Description: The surgeon will complete an assessment of the following:
  1. Closure Method Satisfaction
  2. Scar Satisfaction
  3. Wound Healing as judged by Wound Evaluation Scale
  Scale rated on 1 (least favorable) to 6 (most favorable)
  Please note that only 18 patients were evaluated (of 19) in the Standard Suture Closure due to one patient withdrawing from the trial.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
units on a scale | 6 (0) | 6 (0)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

5. Secondary Outcome: Surgeon Satisfaction With Scar
Description: At 3 months post-procedure, the surgeon evaluated their satisfaction on a scale from 1 to 5, 5 being the least favorable.
  Please note that only 18 patients were evaluated (of 19) in the Standard Suture Closure due to one patient withdrawing from the trial.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
units on a scale | 1 (0) | 1.06 (0.24)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.462, t-test, 2 sided

6. Secondary Outcome: Patient Comfort
Description: At 2 weeks post-procedure, patient comfort was evaluated with a scale 1 (most favorable) to 5 (least favorable).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 19
units on a scale | 1.77 (1.15) | 1.94 (1.16)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.646, t-test, 2 sided

7. Secondary Outcome: Patient Satisfaction With Scar
Description: Patient will complete questionnaires that includes assessments of the following:
  1. Pain
  2. Closure Method Comfort
  3. Closure Method Satisfaction
  4. Scar Satisfaction
  Scar Satisfaction was measured on a scale from 1 (most satisfied) to 5 (least satisfied)
  Please note that only 18 patients were evaluated (of 19) in the Standard Suture Closure due to one patient withdrawing from the trial.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
units on a scale | 1.32 (0.48) | 1.22 (0.43)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.510, t-test, 2 sided

8. Secondary Outcome: Patient Rating of Scar
Description: At 3 months post-procedure, patients were asked to rate their scar. Scale was measured from 0 (best scar) - 10 (worst scar)
  Please note that only 18 patients were evaluated (of 19) in the Standard Suture Closure due to one patient withdrawing from the trial.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
units on a scale | 0.87 (0.76) | 1.04 (1.39)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.651, t-test, 2 sided

9. Secondary Outcome: Patient Incision Pain
Description: At the discharge visit, patients evaluated their level of pain at the incision site based on a scale 1 (least pain) through 10 (worst pain).
Time Frame: 1 day (discharge)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 19
units on a scale | 1.77 (2.48) | 2.15 (1.83)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.588, t-test, 2 sided

10. Secondary Outcome: Patient Incision Pain
Description: At 2 week post-procedure, incision pain was evaluated on a scale 0 to 10 (worst pain).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 19
units on a scale | 0.64 (0.92) | 0.71 (1.41)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 0.858, t-test, 2 sided

11. Secondary Outcome: Patient Incision Pain
Description: Incision pain experienced by the patient was evaluated at 3 months post-procedure. This was evaluated on a scale of 0 (least pain) to 10 (worst pain).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Number analyzed (Participants) | 21 | 18
units on a scale | 0.27 (0.41) | 0.27 (0.73)
Statistical Analysis 1: Comparison: Zip Surgical Skin Closure Device vs Standard Suture Closure; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Zip Surgical Skin Closure Device | Standard Suture Closure
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No